CLINICAL TRIAL: NCT04412772
Title: A Randomized, Controlled Clinical Trial of the Safety and Efficacy of Tocilizumab for the Treatment of Severe COVID-19
Brief Title: Trial of Tocilizumab for Treatment of Severe COVID-19: ARCHITECTS
Acronym: ARCHITECTS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per Queen's Regulatory Office, study is terminated or expired.
Sponsor: Queen's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA-2020-019
Record Dates: First submitted 2020-06-01; First posted 2020-06-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tocilizumab (TCZ) Arm (Experimental): Participants will receive 1 intravenous (IV) infusion of TCZ, dosed at 8 mg/kg, up to a maximum dose 800 mg. Up to 1 additional dose may be given if clinical symptoms worsen.
  Interventions: Drug: Tocilizumab
- Placebo Arm (Placebo Comparator): Participants will receive 1 IV infusion of placebo matched to TCZ. Up to 1 additional dose may be given if clinical symptoms worsen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive 1 dose of IV TCZ. 1 additional dose may be given if clinical symptoms worsen.
  Other Names: Actemra
  Arms: Tocilizumab (TCZ) Arm
Drug: Placebo — Participants will receive 1 dose of IV placebo matched to TCZ. Up to 1 additional dose may be given if clinical symptoms worsen.
  Arms: Placebo Arm

SUMMARY:
The overall objective is to evaluate the clinical efficacy and safety of tocilizumab relative to placebo among approximately 300 hospitalized adult patients who have severe COVID-19. The study will be a 2 arm double blinded comparison between tocilizumab 8 mg/kg and matching placebo IV. The dose may be repeated in 8-12 hours if clinical symptoms worsens, (e.g. increase in oxygen requirements). Participants will be followed for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* ii. Hospitalized with COVID-19 pneumonia, based on chest X-ray or CT scan AND iii. Evidence of hyperinflammation: IL-6>40pg/mL (if available) OR CRP >2 mg/dL OR ferritin >2000 ng/mL AND iv. One or more of the following: impending need for requiring invasive or non-invasive mechanical ventilation OR shock requiring vasopressor (without evidence of bacterial / fungal infection) OR need for extracorporeal membrane oxygenation (ECMO) OR severe, refractor ARDS (PaO2/FiO2<200 mmHg)

Exclusion Criteria:

Known severe allergic reactions to tocilizumab or other monoclonal antibodies

* Active tuberculosis infection based on history
* Suspected active bacterial, fungal, viral, or other infection (besides COVID-19)
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Have received oral anti-rejection or immunomodulatory drugs (including tocilizumab) with the past 6 months
* Participating in other drug clinical trials (participation in COVID-19 trials allowed)
* Self-reported pregnant or breastfeeding
* Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 10 x upper limit of normal (ULN) detected within 24 hours at baseline
* Absolute neutrophil count (ANC) < 1000/mL at baseline
* Platelet count < 50,000/mL at baseline

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical status (on a 7-point ordinal scale) at day 28 | up to day 28
  Clinical Status 7-point ordinal scale:
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or ECMO
  7. Death

SECONDARY OUTCOMES:
Clinical improvement | up to day 28
  ii. Time to clinical improvement, defined as a National Early Warning Score (NEWS) of < 2 maintained for 24 hours iii. Time to clinical improvement of at least 2 categories relative to baseline on a 7-category ordinal scale of clinical status
Mechanical Ventilation | up to day 28
  iv. Incidence of mechanical ventilation v. Ventilator-free days
Oxygenation | up to day 28
  vi. Duration of time on supplemental oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Todd Seto, MD, Principal Investigator — The Queen's Medical Center
Locations (1):
- Queen's Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No